CLINICAL TRIAL: NCT04889937
Title: A Study to Evaluate the Usability, Adherence and Diagnostic Performance of a Novel System to Non-Invasively Detect Severe Neutropenia
Brief Title: Usability, Adherence and Diagnostic Performance of PointCheck in Pediatric Population
Acronym: PC004
Status: Completed | Type: Observational
Sponsor: Leuko Labs, Inc. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other); Center for Advancing Point of Care Technologies (Other)
Responsible Party: Sponsor
Other Study IDs: MDACC Protocol ID: 2021-0061
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PC004 Cohort: The study will include a sample of patients with specific cancer types visiting the outpatient hematologic oncology clinic for their standard of care chemotherapy administration. Participants will need to be willing to participate and be able to provide written informed consent
  Interventions: Device: PointCheck

INTERVENTIONS:
Device: PointCheck — PointCheckTM is intended for use to aid in the assessment of severe neutropenia in the home or clinic setting in subjects receiving myelosuppressive chemotherapy with intermediate to high febrile neutropenia risk. The device non-invasively captures real-time videos of blood flow in the nailfold microcirculation and utilizes visible light, a microscope and a computer vision software to provide a qualitative result. The device is limited to use as a preliminary assessment tool in conjunction with standard of care, including temperature monitoring and clinical assessment. It is not to be used as a stand-alone determinant of severe neutropenia or for any other diagnostic purpose

SUMMARY:
Single-site non-significant risk, open-label clinical investigation designed to validate the usability, adherence, and preliminary diagnostic performance of a novel technology to detect neutropenia. Study participants will be managed as per the standard of care practice with a baseline and nadir visit including laboratory determinations. Participants will also be evaluated with the device at both time points and with daily measurements during the two-week period in between.

ELIGIBILITY:
Inclusion Criteria

1. Study subjects, or their parent/legal guardian for subjects <18 years, must be able to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local subject privacy regulations. Subjects between the ages of 7 and 17.9 years must provide assent.
2. Male or Female aged 7 years to 65 years.
3. Adults (> 18 years) diagnosed Diagnosed with Hodgkin/Non-Hodgkin Lymphoma or breast cancer.
4. Children and adolescents (7 - 18 years) with liquid or solid tumors.
5. Scheduled treatment with cytotoxic chemotherapy with an associated high/intermediate risk of neutropenia (table 1) 30.
6. Able (in the investigator's opinion) and willing to comply with all study requirements.

Exclusion Criteria

1. Participants with amputations, congenital malformations, or any severe abnormalities of the hands as determined by the investigator.
2. Participants with a history of vasculitis, Raynaud syndrome, scleroderma, mixed connective tissue disease, or any other rheumatologic systemic condition that could produce microcirculatory changes in the nailfold.
3. Participants with circulating tumor cells in previous or current lab determinations.
4. Adult (>18 years) participants with leukemia of all types and pediatric (7-18 years) participants with leukemia that are either not in remission or in the minimal residual disease category.
5. Participants with any condition producing significant tremor (e.g., essential tremor, Parkinson´s disease, dystonic tremor).
6. Unstable participants (pediatric or adults) or adult participants with hypotension (systolic blood pressure <90 and diastolic blood pressure < 60mmHg).
7. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
8. Other unspecified reasons that, in the opinion of the Investigator or Sponsor, make the subject unsuitable for enrolment.

Ages: 7 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will be conducted in children, and adults diagnosed with cancer that require cytotoxic chemotherapies that could lead to febrile neutropenia. Patients with Diffuse Large B-Cell Non-Hodgkin Lymphoma (DLBCL) and breast cancer who are scheduled to receive cytotoxic chemotherapy agents with high (>20%) or intermediate (10-20%) risk of neutropenia will be the main target. However, all adult patients with Hodgkin/Non-Hodgkin Lymphoma and breast cancer and all children with solid or liquid tumors (see inclusion and exclusion criteria) whose therapy has an intermediate or high-risk of febrile neutropenia, are eligible. The main factor to select the populations will therefore be the estimated risk of severe neutropenia from the chemotherapy used. Patients under any other regimen that have an associated FN risk greater than 10% will be considered eligible.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Usability of PointCheck | Up to three-weeks
  The study will confirm if participants can acquire good quality videos in a home like setting.
  The System Usability Scale (0-100 higher scored indicate a better usability) will be completed by the participants after completing the follow up visit.

SECONDARY OUTCOMES:
Accuracy of PointCheck | Up to three-weeks
  The preliminary diagnostic accuracy to detect grade IV neutropenia according to CTCAE V5 (<500 ANC/mm3) measured by the sensitivity and the specificity will be the evaluated with reference to the corresponding laboratory measures acquired at the nadir (follow up) visit.
Repeatability of PointCheck | Up to three-weeks
  The % agreement of the device to classify neutropenia compared to the laboratory reference will be established
Number of participants with device-related adverse events as assessed by CTCAE v5.0 | Up to three-weeks
  The number (and %) of AEs, SAEs and their relationship with the device use will be the safety endpoint
Adherence to PointCheck | Up to three-weeks
  The number of days that the participant used the device will be used to evaluate adherence.

OTHER OUTCOMES:
Predictive capacity of PointCheck | Up to three-weeks
  An exploratory analysis about the number of days before the second lab determination that PointCheckTM detected severe neutropenia will be investigated in those participants with severe neutropenia at the nadir visit. Also, exploratory analysis will be conducted in patients developing febrile neutropenia (axillary temperature ≥100.4°F and grade III/IV neutropenia documented in the lab report) during the study to evaluate how many days before the appearance of fever the device detected severe neutropenia during the at home phase of the study.
Diagnostic performance for a second cutoff | Up to three-weeks
  The preliminary diagnostic accuracy to detect grade III neutropenia according to CTCAE V5 (<1000 ANC/mm3) 13 measured by the sensitivity and the specificity will be the evaluated with reference to the corresponding laboratory measures acquired at the nadir (follow up) visit.
Clinical Utility Assessment | Up to three-weeks
  Survey completed by the clinical team at the baseline visit assessing the clinical utility of PointCheckTM

CONTACTS AND LOCATIONS:
Overall Officials: Branko Cuglievan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- See also: Sponsor website — https://leuko.com/